CLINICAL TRIAL: NCT01145794
Title: Reducing Secondhand Smoke Exposure Among Young Children in Shanghai, China
Brief Title: Secondhand Smoke Exposure Reduction Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: Flight Attendant Medical Research Institute (Other)
Responsible Party: Abu Abdullah/Associate Professor, Boston University School of Public Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: China-SHARE
Record Dates: First submitted 2010-06-15; First posted 2010-06-17 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Secondhand Smoking
Keywords: SHS

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: smoking hygiene intervention — The intervention, SHI, will address SHS and quitting. It will include behavioral counseling to address health hazards of SHS for children, brief advice to quit and to adopt a no smoking policy around children and self-help materials (related to second hand smoking).

SUMMARY:
The high prevalence of smoking in adults in many developing countries (e.g. in China, 61% among men and 7% among women) results in many children being exposed to secondhand smoke (SHS). Although in 2001 the American Academy of Pediatrics recommended the promotion of proper smoking hygiene, (i.e. smoking away from the immediate environment of infants and children), similar recommendations in many developing countries are either scarce or non-existent. We hypothesize that implementation of a package of smoking hygiene intervention measures delivered by community health workers (CHWs) will reduce Chinese children's exposure to SHS and improve their respiratory health.

ELIGIBILITY:
Inclusion Criteria:

1. household member has smoked one or more cigarettes daily for the past 30 days as self reported;
2. household smoker smokes a total of at least 10 cigarettes per week at home in the presence of the child, as self reported;
3. smoker household member and the child are living together in the same household and will live together during the entire period of the study;
4. residents of the study community;
5. able to communicate in Mandarin Chinese or local Shanghai dialect;
6. has signed an informed consent form or given verbal consent (for those who cannot read and write).

Exclusion Criteria:

1. reported residential coal burning and confirmed by the interviewer;
2. households with breast-feeding child;
3. household members do not smoke at home;
4. smoker member does not live in the same household as the under 5 child;
5. non-local community resident; and
6. not able to communicate in Mandarin Chinese or Shanghai dialect.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 348 (Estimated)
Dates: Start 2008-10; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
improvement of smoking hygiene practices within the household as reported by the subjects | at 6 months
  The main outcome measures are: improvement of smoking hygiene practices within the household as reported by the subjects (i.e. reduction in the number of cigarettes smoked indoors at home while a child was present during the previous week) and reduction in children's cotinine concentrations in urine at 6- month follow up.

CONTACTS AND LOCATIONS:
Locations (1):
- Fu Hua, Shanghai, China